CLINICAL TRIAL: NCT06169787
Title: Sentinel Lymph Nodes Biopsy Versus Lymphadenectomy in Cervical Cancer
Brief Title: Sentinel Lymph Nodes Biopsy in Cervical Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Professor, Far Eastern Memorial Hospital
Other Study IDs: 112154-E
Record Dates: First submitted 2023-10-14; First posted 2023-12-14 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-04

CONDITIONS: Sentinel Lymph Node
MeSH Terms: interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sentinel Lymph Node: Sentinel lymph node biopsy in patients with early stage cervical cancer
  Interventions: Procedure: sentinel lymph node biopsy
- Lymphadenectomy: Comprehensive lymphadenectomy in patients with early stage cervical cancer
  Interventions: Procedure: comprehensive pelvic lymphadenectomy

INTERVENTIONS:
Procedure: sentinel lymph node biopsy — sentinel lymph node biopsy
  Groups: Sentinel Lymph Node
Procedure: comprehensive pelvic lymphadenectomy — comprehensive pelvic lymphadenectomy
  Groups: Lymphadenectomy

SUMMARY:
This study aims to compare sentinel lymph nodes biopsy versus comprehensive lymphadenectomy in patients with early stage cervical cancer who underwent radical hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

Women aged 20 and above with clinical FIGO stage I-IIA cervical cancer

Exclusion Criteria:

Women did not receive surgical treatment

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with early stage cervical cancer
Study Population: Women aged 20 and above with early stage cervical cancer, who received surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-10-14 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 5 years
  progression free survival between these two groups

SECONDARY OUTCOMES:
overall survival | 5 years
  overall survival between these two groups
Number of dissected lymph node | 5 years
  Number of dissected lymph node between these two groups

OTHER OUTCOMES:
Complications | 5 years
  Compication rates between the traditional and sentinel lymph node dissection groups

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No